CLINICAL TRIAL: NCT05674201
Title: Effects Of Propofol-Dexmedetomıdıne And Propofol- Remıfentanıl On Recovery And Hemodynamıcs In Hysteroscopıc Operations, That One Of The Ambulatory Anesthesıa Practices: A Randomızed Controlled Study
Brief Title: Effects Of Propofol-Dexmedetomıdıne And Propofol- Remıfentanıl In Hysteroscopıc Operations.
Status: Completed | Type: Observational
Sponsor: Siirt Training and Research Hospital (Other Government)
Collaborators: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, ali kendal oğuz, medical doctor, Siirt Training and Research Hospital
Other Study IDs: SiirtTRH
Record Dates: First submitted 2022-12-07; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Deep Sedation; Ambulatory Surgery; Ambulatory Surgical Procedure
Keywords: Ambulatory Anesthesia; Hysteroscopy; Sedation; Dexmedetomidine; Remifentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Group DP: Propofol (Dexmedetomidine (Sedadomide 200 µg/2 ml, KOÇAK FARMA Turkey)
  1mcg/kg bolus was administered to Group DP in 10 minutes, then 0.2-1.4 mcg/kg/hour infusion dose was started.-®Lipuro 1%(10 mg/ml), B. Braun Indonesia ) 1mg/kg bolus was administered.
  Interventions: Combination Product: Propofol-Dexmedetomidine
- Group RP: Propofol (Propofol-®Lipuro 1%(10 mg/ml), B. Braun Indonesia ) 1mg/kg bolus was administered, After a 0.25mcg/kg bolus of Remifentanil (Ultiva®, GlaxoSmithKline, Belgium) was administered to Group RP, a 0.025-0.1mcg/kg/minute infusion dose was started.
  Interventions: Combination Product: Propofol-Dexmedetomidine

INTERVENTIONS:
Combination Product: Propofol-Dexmedetomidine — Propofol-Dexmedetomidine AND Propofol-Remifentanil
  Other Names: Propofol-Remifentanil

SUMMARY:
In our study, the investigators aimed to compare the effects of dexmedetomidine-propofol and remifentanil-propofol combinations on perioperative spontaneous respiration, hemodynamics, recovery, participants, surgeon and anesthetist satisfaction in hysteroscopy, which is one of the ambulatory surgery.

DETAILED DESCRIPTION:
This study was conducted prospectively after the approval of Van Yüzüncü Yıl University Ethics Committee. A total of 80 participants in 2 groups of 40 ASA I-II, aged 18-65 years were included in the study. On the day of the operation, vascular access was established with a 20 G branule in all patients before the procedure. The participants who were taken to the gynecology table were routinely monitored in the supine position as required by the procedure.

All participants were premedicated with 0.025 mg/kg Midazolam (Demizolam®, Dem, Turkey) after starting oxygen at 2 lt/min with a nasal cannula. The participants were randomly divided into two groups as Group DP and RP. Propofol (Propofol-®Lipuro 1%(10 mg/ml), B. Braun Indonesia ) 1mg/kg bolus was administered to both groups. Dexmedetomidine (Sedadomide 200 µg/2 ml, KOÇAK FARMA Turkey)

1mcg/kg bolus was administered to Group DP in 10 minutes, then 0.2-1.4 mcg/kg/hour infusion dose was started. After a 0.25mcg/kg bolus of Remifentanil (Ultiva®, GlaxoSmithKline, Belgium) was administered to Group RP, a 0.025-0.1mcg/kg/minute infusion dose was started.Hemodynamic data and respiratory parameters of the groups before and after sedation were recorded. The depth of anesthesia was recorded using the Ramsey sedation scale, and the recovery scores were recorded with the Modified Aldrete score. The facial pain scale was used to evaluate pain. Depth of anesthesia was provided so that the Ramsey Sedation Scale of the patients was greater than four. Patients with RSS<4 were excluded from the study by administering additional propofol.

ELIGIBILITY:
Inclusion Criteria:

AGE 18-65 ASA I AND II

Exclusion Criteria:

* OTHERS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted prospectively after the approval of Van Yüzüncü Yıl University Ethics Committee. A total of 80 patients in 2 groups of 40 ASA I-II, aged 18-65 years were included in the study.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
SEDATİON | through study completion, an average of 1 year
  RAMSEY SEDATİON SKORE > 4 TİME (MİNUTE)
RECOVERY | through study completion, an average of 1 year
  MODIFIED ALDRETE SCORE>9 (MİNUTE)
DESATURATION DESATURATION | DURING THE SURGERY
  SATURATION SATURATION RATIOS (%)
RESPİRATORY RATE | DURING THE SURGERY
  RESPİRATORY RATE (.../MİNUTE)
END-TİDAL CO2 | DURING THE SURGERY
  END-TİDAL CO2 (mmHg)
INTEGRATED PULMONARY INDEX | DURING THE SURGERY
  INTEGRATED PULMONARY INDEX (1-10)

SECONDARY OUTCOMES:
HEART RATE | DURING THE SURGERY
  HEART RATE (../MİNUTE)
NON INVASIVE SYSTOLİC AND BLOOD PRESSURE | DURING THE SURGERY
  NON INVASIVE BLOOD PRESSURE ( mmHg)
NON INVASIVE DİASTOLİC BLOOD PRESSURE | DURING THE SURGERY
  NON INVASIVE BLOOD PRESSURE ( mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Siirt Eğitim Ve Araştirma Hastanesi, Siirt, Turkey (Türkiye)

REFERENCES:
- [Derived] Oguz AK, Soyalp C, Tuncdemir YE, Tekeli AE, Yuzkat N. Sedoanalgesia with dexmedetomidine in daily anesthesia practices: a prospective randomized controlled trial. BMC Anesthesiol. 2025 Jan 29;25(1):45. doi: 10.1186/s12871-025-02918-1. PMID 39881245